# **Proprietary Information of MD Anderson**

2018-0489 PI: Amin Alousi NCT ID: NCT04239989

Informed Consent Document March 27, 2023



#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

A Phase I Study to Assess Safety of Selective JAK 1 Inhibitor, Itacitinib, in Patients with Bronchiolitis Obliterans syndrome (BOS) after Allogeneic Hematopoietic Cell Transplant (HCT) 2018-0489

| Study Chair: | Amin Majid Alousi |
|--------------------|-----------------------|
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB – a committee that reviews research studies).

# STUDY SUMMARY

The goal of this clinical research study is to learn if itacitinib is safe to give to patients who have bronchiolitis obliterans syndrome (BOS) after having received an allogeneic stem cell transplant. Researchers also want to find out if itacitinib may relieve the symptoms of BOS.

**This is an investigational study.** Itacitinib is not FDA approved or commercially available. Its use in this study is for research purposes only. The study doctor can explain how the study drug is designed to work.

Treatment with the study drug may help to control BOS. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

You can read a list of potential side effects below in the Possible Risks section of this consent.

Itacitinib and the bronchoscopy performed at screening and at 6 months will be provided at no cost to you while on this study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive the standard-of-care treatment for BOS such as steroids and/or immune system suppressing drugs. The study doctor will discuss the standard treatments available to you, including their risks and benefits. You may choose to receive other investigational therapy, if available. You may choose not to have treatment for BOS at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of BOS.

#### 1. STUDY DETAILS

# **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible. If you have had some of these tests recently, they may not need to be repeated.

- You will have a physical exam.
- Blood (about 2 teaspoons) will be drawn for routine tests, to check your thyroid function, and to test for infectious diseases, such as human immunodeficiency virus (HIV), and a separate test for tuberculosis (TB). If you can become pregnant, part of the blood will be used for a pregnancy test. To take part in this study, you cannot be pregnant.
- You will have lung function tests.
- If you speak English, you will complete 4 questionnaires about your symptoms and ability to breathe. They should take about 10-20 minutes to complete.
- You will complete a 6-minute walk test.
- You will have a bronchoscopy to collect samples of fluid from your lungs to check the status of your disease and for biomarker testing. Your doctor will explain how this test is done. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug. Biomarker testing is being done for research purposes only, and the results will not be used to decide if you are eligible to take part in this study. You will sign a separate bronchoscopy consent that describes this procedure and its risks in more detail.
- You will have CT scans of your chest as part of standard of care to check the status of your disease.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in this study, you will not be enrolled. Other options will be discussed with you.

Up to 15 patients will enrolled in this study. All will take part at MD Anderson.

# **Study Drug Administration**

Each study cycle is 28 days.

If you are found eligible to take part in this study, you will take itacitinib (2 tablets) by mouth 1 time a day on Days 1-28 of each cycle for up to 1 year. Itacitinib may be taken with or without meals.

You will receive prednisone by mouth every day for 2 weeks to help decrease the risk of side effects. After 2 weeks, you will slowly start to take lower doses of prednisone, until your doctor thinks you no longer need to take it. Your doctor will explain how many tablets to take each day.

You should bring any unused study drug to the clinic to dispose of it at each study visit. You can also dispose of the drug at home. The study staff will give you instructions for how to do this.

You will also receive a pill diary in which you will record when you take each dose. The study staff will give you instructions for this as well.

# **Study Visits**

At Week 1, Week 2, and then once a month from Months 1 through 13, blood (about 2 teaspoons) will be drawn for routine tests. If you can become pregnant, part of the blood sample or a urine sample will be collected for a pregnancy test. To continue taking part in this study, you cannot be pregnant.

#### At 3 months and 6 months:

- You will have lung function tests.
- If you speak English, you will complete the 4 questionnaires you completed at screening.
- You will complete a 6-minute walk test.

#### At 6 months:

- You will have a bronchoscopy to collect samples from your lungs to check the status of your disease and for biomarker testing. You will sign a separate consent for this procedure.
- You will have CT scans as part of standard of care to check the status of your disease.

At **12 months**, you will have lung function tests.

You will also have other standard of care tests to check the status of the disease during the study. Outside laboratory visits can be done at Week 1 and Week 2, and then at Months 1, 2, 4, 5, and 7-11.

#### Other Information

While taking itacitinib, avoid having any grapefruit and pomegranate juice or other products containing grapefruit or pomegranate.

You cannot receive any other anticancer or investigational therapy or a JAK inhibitor (drugs similar to Itacitinib) while you are taking the study drug.

If you need to use aspirin or aspirin-containing medications, use them with caution. You should discuss this with the study doctor.

Ask the study doctor before taking any other drugs, since they may interfere with the study drug.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting, or permanent, and may even result in hospitalization and/or death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drug.

# **Itacitinib Side Effects**

This is an early study of itacitinib in humans, so the side effects are not well known. Based on studies in early studies in humans, itacitinib may cause the following side effects:

# Common (occurring in more than 20% of patients)

| fatigue | diarrhea | low blood cell counts |
|---------|--------------------------|-------------------------|
| | <ul><li>nausea</li></ul> | (red, platelets, white) |

Itacitinib may cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue.
   You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere, such as your mouth or urinary tract, and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# Occasional (occurring in 3-20% of patients)

| • | fever due to a low white | weakness | <ul> <li>severe life-threatening</li> </ul> |
|---|---|---|---|
| | blood cell count | | infection (which may |
| • | vomiting | | lead to low blood |
| | • | | pressure, kidney failure, |
| | | | and/or heart failure) |

There are currently no known side effects occurring in fewer than 3% of patients.

# **Prednisone Side Effects**

# It is not known how often the side effects of prednisone may occur:

- heart failure
- high blood pressure
- swelling
- headache
- increased pressure between the skull and brain (possible swelling of the eye nerve, vision changes, and/or headaches)
- mental health disturbances (including euphoria [unusual feelings of happiness or well-being])
- difficulty sleeping
- mood swings
- personality changes
- severe depression
- seizure
- fatigue and anxiety
- dizziness
- bruising
- facial skin redness
- tiny dots on the skin
- thin fragile skin
- hives
- sweating
- wound healing problems
- Cushing's syndrome (possible weakness, diabetes, and/or bone weakness)

- failure of hormoneproducing organs
- decreased ability to process carbohydrates
- high level of steroid in the body (possible mood changes and diabetes)
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)
- diabetes
- abnormal blood acid/base balance (possible organ damage)
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- body-wide loss of proteins (possible weakness and/or swelling)
- low blood levels of potassium (possible muscle cramps)
- high blood levels of sodium (possible weakness and/or swelling)
- abdominal swelling
- inflammation of the pancreas (possible

- stomach ulcer (with possible hole and bleeding)
- esophagus sore
- abnormal liver or bone tests (possible liver damage)
- pain or loss of function of the hips and/or shoulders due to bone death
- loss of muscle
- muscle weakness (possibly caused by muscle damage)
- loss of bone strength (possible broken bones)
- brittle/broken bones
- tendon tear (particularly Achilles tendon)
- collapse of bones in the spine
- bulging eye
- increased pressure in the eye (possible vision loss, pain, and/or blurry vision)
- cataracts (clouding of the lens of the eye)
- allergic reactions that are possibly lifethreatening (such as difficulty breathing, low blood pressure, and/or organ failure)

| abdominal pain) |
|-----------------|

# Rarely (in fewer than 3% of patients)

• blood clots in a vein (possible pain, swelling, and/or redness)

Prednisone may cause an increased risk of infection, such as pneumonia. This infection may occur anywhere. It may become life-threatening. Symptoms of infection may include fever, pain, redness, and/or difficulty breathing.

Prednisone may cause you to develop another type of cancer (such as Kaposi's sarcoma).

#### **Other Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**Bronchoalveolar lavage** may cause cough, fever, chills, and/or muscle pain. It may cause difficulty breathing due to narrowing of the airways. You may need a ventilator to help you breathe.

It is not known how often the following side effects of **bronchoscopy** may occur.

| <ul> <li>irregular heartbeat</li> <li>chest pain</li> <li>fever</li> <li>bleeding</li> <li>low oxygen level in the blood (possible lightheadedness)</li> </ul> | <ul> <li>collapsed lung (possible difficulty breathing)</li> <li>possible need for a breathing tube</li> <li>sore throat</li> </ul> | <ul> <li>cough</li> <li>difficulty breathing<br/>(possibly due to<br/>narrowing of the<br/>airways)</li> <li>blood in the mucus</li> </ul> |
|---|---|---|
|---|---|---|

Bronchoscopy may cause an increased risk of infection, such as pneumonia. This infection may occur anywhere. It may become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

You may have stinging, burning, tingling, and/or tenderness of the mouth and/or difficulty swallowing when you gargle with the anesthetic before the procedure.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.

**Lung function tests** may cause dizziness and/or fainting. If you feel lightheaded, tell the study doctor or study team. For people with asthma, the test may cause an asthma attack. In very rare cases, lung function tests may cause a collapsed lung.

**CT scans** send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study. Only authorized people who are working on this study will have access to study data

This study may involve unpredictable risks to the participants.

# **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you are able to become pregnant or father a child, you must use appropriate birth control while you are on study. Talk to the study staff about appropriate methods of birth control.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant may result in your removal from this study.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Incyte, Ltd. for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- 4. You may ask the study chair (Dr. Amin Alousi, at 713-745-8613) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can help you safely stop study treatment. It may be dangerous to suddenly stop study treatment. The study doctor will also decide if you need to have any visits or tests to check on your health. If you withdraw from this study, you can still choose to be treated at MD Anderson.
  - If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can continue to collect data from your routine medical care. If you agree, this data will be handled the same as research data.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Incyte, Ltd., the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.

- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
  - Most tests done on samples in research studies are only for research and have no clear meaning for health care. If the research with your identifiable information or samples gives results that do have meaning for your health, the researchers will contact you to let you know what they have found.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is supported by: Incyte, Ltd
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

Your personal information and/or samples are being collected as part of this study. These data and/or samples may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

Before being shared for future research, every effort will be made to remove your identifying information from any data and/or samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or samples are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples or data at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### Genetic Research

Samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

#### **Outside Care**

Part of your care may be provided outside of MD Anderson by your home doctor(s).

#### **Conflict of Interest**

Dr. Amin Alousi (Study -Chair) has received compensation from Incyte as a Consultant. The financial interests are within the limits of the conflict of interest policy.

# Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson

- Incyte, Ltd, who is a supporter of this study, and/or any future sponsors/supporters of the study
- Any future sponsors and/or licensees of the study technology
- Study monitors and auditors who verify the accuracy of the information
- Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performed | under this protocol. |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| I have discussed this research study with the participant and/or his or representative, using language that is understandable and appropriat have fully informed this participant of the nature of this study and its pand risks and that the participant understood this explanation. | e. I believe that I possible benefits |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |
| TRANSLATOR I have translated the above informed consent as written (without addi subtractions) into and assisted to (Name of Language) obtaining and providing consent by translating all questions and responsent process for this participant. | the people |
| NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR | DATE |
| ☐ Please check here if the translator was a member of the research a witness, other than the translator, must sign the witness line.) | team. (If checked, |

Photocopies Allowed After Signatures Obtained Edited IRB Activated Consent/Authorization , Date of Consent Activation: 4/12/2023